CLINICAL TRIAL: NCT01516242
Title: Monitoring of Expected Parameters of the Application Technique and Safety of the Therapy
Brief Title: Evaluation of Safety and Parameters of Application Technique
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: MS236-1926
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NovoPen® 4
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Collection of data about patients with type 1 diabetes or type 2 diabetes treated with insulin changing their insulin administration from syringe to a insulin delivery system based on completion of questionaire

SUMMARY:
This study is conducted in Europe. The aim of the study is to monitor patients changing therapy from syringe to insulin delivery system as prescribed by the treating physician in Slovakia.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (type 1 or type 2)
* Treated with insulin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 1 diabetes or type 2 diabetes mellitus treated with insulin having changed administration of inulin from syringe to a Novo Nordisk insulin delivery system
Sampling Method: Probability Sample
Enrollment: 4819 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Number of insulin applications (punctures)
Reasons leading to change of the therapy
Patient satisfaction with NovoPen® 4 insulin delivery system

SECONDARY OUTCOMES:
Adverse reactions
Hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bratislava, Slovakia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com